CLINICAL TRIAL: NCT03035877
Title: Treatment of Justice-Involved Emerging Adults With Substance Use Disorders
Brief Title: Multisystemic Therapy-Emerging Adults (MST-EA) for Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: University of Massachusetts, Worcester (Other); Connecticut Department of Children and Families (Unknown); North American Family Institute (Unknown); Court Support Services Division (Unknown); Youth Villages (Other); Chestnut Health Systems (Other)
Responsible Party: Principal Investigator, Ashli Sheidow, Senior Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DA041425-01 (NIH)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Antisocial Behavior
Keywords: Antisocial Behavior; Alcohol Abuse; Drug Abuse; Young Adults
MeSH Terms: conditions — Antisocial Personality Disorder; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisystemic Therapy-Emerging Adults (Experimental): This group will receive Multisystemic Therapy-Emerging Adults.
  Interventions: Behavioral: Multisystemic Therapy-Emerging Adults
- Enhanced Treatment as Usual (Active Comparator): This group will have access to an enhanced version of services typically delivered to young adults who have a substance use disorder and have been in trouble with the law.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Multisystemic Therapy-Emerging Adults — MST-EA is a home- and community-based treatment for emerging adults (ages 17-21) that aims to address antisocial behavior and problems caused by substance use disorders. The model also addresses co-occurring mental health problems when present. Therapists work directly with the young adult and his/her social network. This treatment also involves the use of coaches who help young people develop skills for young adulthood.
  Other Names: MST-EA
  Arms: Multisystemic Therapy-Emerging Adults
Behavioral: Enhanced Treatment as Usual — With Enhanced Treatment as Usual (E-TAU), emerging adults will get the treatments that they usually receive when they have a substance use disorder and have been in trouble with the law. In addition, they will receive travel vouchers for attending services, a card with an individualized list of contacts when in crisis, and facilitation with identifying need of services and accessing those services.
  Other Names: E-TAU
  Arms: Enhanced Treatment as Usual

SUMMARY:
This study's purpose is to examine the effectiveness of a promising intervention for emerging adults (EAs) with alcohol and other drug (AOD) abuse and justice involvement in achieving the ultimate outcome of reduced criminal activity. The study will also examine that effect on intermediate outcomes as follows: 1) reduced AOD use; 2) greater gainful activity (increased educational success, employment and housing stability; decreased antisocial peer involvement and relationship conflict); 3) and greater improvement in self-regulation (self-efficacy, goal directedness and responsibility taking). The intervention to be tested is Multisystemic Therapy-Emerging Adults (MST-EA). MST-EA is an adaptation of MST, a well-established, effective intervention for antisocial behavior in adolescents.

DETAILED DESCRIPTION:
Prevalence of alcohol and other drug (AOD) abuse and criminal activity is highest during emerging adulthood compared to any other developmental period, and causes extraordinary costs to society. Emerging Adults (EAs; ages 17-26) with AOD abuse have greater incarceration rates than EAs without AOD abuse, and AOD-abusing offenders have significantly more recidivism, severe offending, and incarceration than other offenders. Such serious behavior interferes with successful transition into adulthood in areas such as school completion, employment and housing. Thus, there is a strong public health need for effective treatment to reduce AOD abuse and justice involvement in EAs. Surprisingly, there are no interventions with established efficacy to reduce criminal activity among EAs, with or without AOD abuse. Among younger adolescents, the comprehensive causes of antisocial behavior are addressed by effective interventions (e.g., Multisystemic Therapy [MST]; Treatment Foster Care Oregon [TFCO]), and the present investigative team has developed and evaluated a well-defined age-tailored intervention for EAs with criminal behavior. The developed intervention is an adaptation of MST and integrates a skills coaching component from TFCO, both well-established effective juvenile justice interventions. Initial MST-EA research focused on justice-involved young adults who had mental health problems, a high-risk subpopulation of offenders, but AOD abuse quickly became a primary problem the MST-EA team treated. As a single-source intervention, MST-EA targets the EA correlates of criminal activity and AOD abuse, including gainful EA activities (positive relationships, school, work, and housing) and reduced AOD abuse-in part by targeting the proximal mechanism of poor self-regulation. In a successfully completed community-based open trial, the safety, feasibility, and preliminary efficacy of the intervention were established.

The proposed study will evaluate the effectiveness of MST-EA for reducing justice involvement and AOD abuse. EAs (n = 240) with AOD abuse and justice involvement (recent arrests or release from justice facilities) will be randomized to receive MST-EA or Enhanced Treatment as Usual (E-TAU). Assessments will be completed at months 0, 2, 4, 6, 8, 12, and 16, with confirmation of outcome data using official records. Aims will be to evaluate the effect over time of MST-EA for reducing AOD abuse and criminal activity, as well as to evaluate the effect of MST-EA on the key proximal target of treatment (self-regulation) and intermediate outcomes of treatment (gainful activities). A final aim of the study will be to investigate if the direct effect of treatment on criminal activity is mediated by its effect on self-regulation, AOD abuse, and gainful activities. In this specific age group, there is a complete absence of AOD abuse and recidivism reduction treatments with demonstrated effectiveness. The ultimate effect of the proposed research would be decreased AOD abuse and justice involvement in a high-risk population, as well as improved outcomes that have significant societal impact (e.g., reduced homelessness and unemployment).

ELIGIBILITY:
Inclusion Criteria:

* Age 16 to 26 years
* Recent arrest or release from jail/prison/detention (within the past 18 months but excluding arrest for parole/probation violations)
* Presence of alcohol or drug (AOD) abuse disorder and recent AOD use (within the past 90 days)
* Able to reside in a stable community setting (not currently homeless, not currently in-patient; can include individuals ready for discharge to the community)

Exclusion Criteria:

* Actively psychotic, suicidal, or homicidal
* Pervasive Development Disorders (PDD) or mental retardation
* Sex offending as the primary offense type

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Change in number and severity of criminal charges in official records in the 16 months pre-Baseline compared with the 16 months post-Baseline. | 16 months pre-Baseline compared with 16 months post-Baseline.
  Changes from the 16 months pre-Baseline in offending as measured by the number and severity of criminal charges in official records compared to 16 months post-Baseline.
Changes from Baseline scores compared to 16 months post-Baseline Offending Behaviors (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Offending behaviors as measured using the Self-Report Offending Scale (self-reports).

SECONDARY OUTCOMES:
Changes from Baseline scores compared to 16 months post-Baseline Self-efficacy (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Self-efficacy as measured using the Self-Efficacy Scale (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline Goal Directedness (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Goal directedness measured using the Wills Self Control Measure (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline Responsibility Taking (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Responsibility taking measured using the Behavioral Indicators of Conscientiousness (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline Urine Drug/Alcohol Screens (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  The number of positive urine screens for tetrahydrocannabinol (THC), synthetic THC, amphetamines, methamphetamines, phencyclidine (PCP), opiates, benzodiazepines, cocaine, and specific metabolites of alcohol (Ethyl glucuronide, Ethyl sulfate).
Changes from Baseline scores compared to 16 months post-Baseline Treatment Usage (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  The number of hospitalizations, emergency room visits and other treatments for alcohol or drug use as measured using the Time Line Follow Back (self-report) and from archival records.
Changes from Baseline scores compared to 16 months post-Baseline Substance Use and Problems (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Frequency of substance use and substance-related problems as measured by the Global Appraisal of Individual Needs (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline Antisocial Peers Involvement (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Antisocial peer involvement measured using the Peer Delinquency Scale (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline Interpersonal Competence (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Social conflict and social functioning as measured using the Interpersonal Competence Scale (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline Housing Stability (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Housing stability as measured using the Time Line Follow Back (self-reports) and from archival records.
Changes from Baseline scores compared to 16 months post-Baseline Relationship Closeness and Discord (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Relational closeness and relational discord as measured by the Network of Relationship Inventory (self-reports).
Changes from Baseline scores compared to 16 months post-Baseline School/Employment Involvement (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  Days in school or work (gainful activities) as measured using the Time Line Follow Back (self-reports) and from archival records.
Changes from Baseline scores compared to 16 months post-Baseline Mental Health Symptoms (measured at 0, 2, 4, 6, 8, 12 and 16 months). | Baseline to 16 months.
  The severity and number of mental health symptoms as measured using the Brief Symptom Inventory and the Posttraumatic Stress Disorder Checklist (self-reports).

CONTACTS AND LOCATIONS:
Overall Officials: Ashli J Sheidow, Ph.D., Principal Investigator — Chestnut Health Systems; Maryann Davis, Ph.D., Principal Investigator — University of Massachusetts, Worcestor
Locations (4):
- United States (4):
  - North American Family Institute, Hamden, Connecticut
  - North American Family Institute, Hartford, Connecticut
  - North American Family Institute, New Haven, Connecticut
  - Youth Villages, Johnson City, Tennessee

IPD SHARING:
Plan to Share IPD: No